CLINICAL TRIAL: NCT03386305
Title: A Randomized Controlled Trial to Evaluate the Clinical Benefits of EnvarsusXR in Post Liver Transplant
Brief Title: Evaluate the Clinical Benefits of EnvarsusXR in Post Liver Transplant
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Albert Einstein Healthcare Network (Other)
Collaborators: Veloxis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Radi Zaki, Co-Chair, Transplantation, Albert Einstein Healthcare Network
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5024
Record Dates: First submitted 2017-12-15; First posted 2017-12-29 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Post Liver Transplant
MeSH Terms: interventions — Immunosuppression Therapy; Tacrolimus; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- EnvarsusXR arm (Experimental): Patients are converted to once daily EnvarsusXR (study drug). The patients continue taking this medication for 9 months of the study. Initial dosage will be 0.8 times the total daily dose of tacro bid, due to higher bioavailability. All subsequent dose adjustments will be based on maintenance of target tacro trough levels within range of 5-12 ng/ml.
  Interventions: Drug: EnvarsusXR
- Standard of care arm (Active Comparator): Post Liver Transplant patients take Tacrolimus twice daily as a part of standard of care. Those participating in the study will continue to take tacrolimus twice daily, as apart of their regular care. As a part of the study, they will complete the medication adherence and quality of life instruments.
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: EnvarsusXR — Patients randomized to study drug will be converted to EnvarsusXR once daily.
  Other Names: Immunosuppression
  Arms: EnvarsusXR arm
Drug: Tacrolimus — Patients continue to take Tacrolimus BID, as a part of routine care.
  Other Names: Standard of Care
  Arms: Standard of care arm

SUMMARY:
This study will evaluate the medication adherence, clinical efficacy, and safety of EnvarsusXR in stable post liver transplant patient using a Phase III randomized controlled study. The primary outcome is change in medication adherence from baseline to the end of the study, assessed using a validated instrument (BAASIS- Basel Assessment of Adherence with Immunosuppressive medication Scales) and standard deviation of Tacrolimus levels.

DETAILED DESCRIPTION:
The main aim of this study is to assess the immunosuppressant adherence, efficacy, and safety in post liver transplant patients converted from twice daily tacro to once daily EnvarsusXR. Tacrolimus trough level, clinical markers of liver disease, HbA1c , eGFR will be assessed at baseline, 1 week, 2 week, 4 week, 3 month and 6 months. Graft rejection will be assessed using routine standard guidelines to identify the cause. All patients post 1 year liver transplant, and within 5 years will be eligible to participate.

The primary hypothesis is that once daily dosing will improve medication adherence in patients randomized to the test arm as compared to the control arm, over a period of 9 months. The clinical efficacy will be assessed by no difference in standard deviation of tacrolimus in the two groups. The secondary hypothesis is that improved medication adherence will lead to improved patient reported quality of life (as assessed by PROMIS-29), and better health outcomes (as assessed by HbA1c, eGFR).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 1 year post liver transplant, but within 5 years of transplant
* Serum Creatinine<= 2.5 mg/dl; AST,ALT, AP and GGT<=2 times ULN
* Patient must be on a stable tacrolimus dose, with tacrolimus trough levels between 5-12 ng/ml for 4 or more weeks before enrolment

Exclusion Criteria:

* Cognitive impairment which precludes participation
* Projected survival, in the opinion of the provider, of less than three months
* Any other solid organ transplant (kidney or pancreas)
* Use of any drug which is known to interfere with tacrolimus metabolism

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2017-12-13 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Medication Adherence | From baseline to 6 months
  Self reported using BAASIS instrument. BAASIS measures taking, skipping and dose reduction of drugs, with a recall period of 4 weeks. It consists of 4 questions with a 6 point response scale (ranging from never to every day). An additional overall adherence is ranked on a scale of 0 to 100 using a visual analog scale.

SECONDARY OUTCOMES:
Change in Quality of life | From baseline to 6 months
  Self reported, using PROMIS-29. PROMIS is a result of the NIH support to develop a "psychometrically validated, dynamic system to measure QOL and patient reported outcomes in study participants. PROMIS-29 comprises a set of 29 questions evaluating seven QOL domains: Physical function, anxiety, depression, fatigue, sleep disturbance, social function and pain. The scores are reported as a T score (mean 50, SD=10) centered on the sample representative of 2000 US general census considering demographic variables.

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Verma, MBBS, MPH, Study Director — Einstein Healthcare Network
Locations (1):
- Einstein Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No